CLINICAL TRIAL: NCT06666816
Title: Observational Study for the Identification of Fatigue and Gait Biomarkers in Populations With Neuromuscular Pathologies in the Clinical Context and Daily Life
Brief Title: Observational Study to Observe Variations of Gait Parameters in Patients With Neuromuscular Diseases
Status: Recruiting | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Other Study IDs: GIP1112; RC 2024-2026 to E. Biffi (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2024-10-25; First posted 2024-10-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Muscular Dystrophies; Myopathies; Spinal Muscular Atrophy (SMA); Charcot Marie Tooth Disease
MeSH Terms: conditions — Muscular Dystrophies; Muscular Diseases; Muscular Atrophy, Spinal; Charcot-Marie-Tooth Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group with neuromuscular disease
  Interventions: Other: inapplicable
- Control Group
  Interventions: Other: inapplicable

INTERVENTIONS:
Other: inapplicable — inapplicable

SUMMARY:
This study has the general objective of observing walking parameters during a clinical test to objectively estimate fatigue in patients with neuromuscular diseases. Furthermore, the investigators want to evaluate the feasibility of collecting physical activity in daily life conditions during a one-week monitoring period using a wearable sensor.

ELIGIBILITY:
Inclusion Criteria:

* Ambulant adult patients with genetic diagnosis of muscular dystrophy/myopathy (dystrophinopathies, muscular dystrophies and congenital and non-congenital myopathies), of spinal muscular atrophy (SMA) and with molecular diagnosis of Charcot-Marie Tooth 1 or 2.
* independent walking, even with assistance;

Exclusion Criteria:

* Dilated or ischemic heart disease with moderate impairment;
* Chronic respiratory failure: forced vital capacity (FVC) < 40%; more than 5% of nocturnal time spent with peripheral oxygen saturation levels < 90.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potentially eligible participants will be selected from clinical databases of IRCCS Medea
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-10-27 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Variation in walking speed during a 6-minutes walking test | Baseline
  Variation in walking speed calculated as difference between the first and the final minute of the a 6-minutes walking test
Subjective fatigue | Baseline
  Evaluation of subjective fatigue using the Fatigue Severity Scale (FSS). The minimum value is 0, the maximum is 63. Higher scores mean worse outcome.

SECONDARY OUTCOMES:
Clinical progression of the neuromuscular disease | Baseline
  Progression of the neuromuscular disease using the Motor Function Measure-32 (MFM-32); the minimum score is 0, the maximum score is 100. Higher values mean better outcome.
Clinical progression of the neuromuscular disease | Baseline
  Progression of the neuromuscular disease using the Hammersmith Functional Motor Scale- Expanded (HFMS-E); the minimum value is 0, the maximum value is 69. Higher values mean better outcome.
Variation in gait variability during the 6-Minutes Walking Test | Baseline
  Variation of step duration during the 6MWT extracted from a wearable inertial sensor. Measured in coefficient of variation (%). Higher values mean worse outcome.

OTHER OUTCOMES:
Acceptability of the activity monitoring device during daily life | Baseline
  Acceptability of the device during activity monitoring in daily life using the Comfort Rating Scale (CRS). Minimum value is 0, maximum value is 20. Higher values mean lower acceptability.
User friendliness of the activity monitoring device during daily life | Baseline
  User friendliness of the device during activity monitoring in daily life using the Questionnaire on User Friendliness of Activity Monitors (QUFAM). Maximum value is 5, minimum value is 0. Higher values mean higher acceptability.
Physical activity in daily life | Baseline
  Steps/day measured using a wearable inertial sensor. Higher values mean better outcome.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Scientific Institute IRCCS E. Medea - Sede di Bosisio Parini, Bosisio Parini, Lecco
  - Scientific Institute IRCCS E. Medea - Polo di Conegliano, Conegliano, Treviso

IPD SHARING:
Plan to Share IPD: Yes
The results obtained at the end of this clinical trial will be presented at national and international conferences and submitted to peer-reviewed international journals. The raw data of the study will be published among the supplementary materials of scientific articles and/or uploaded to Zenodo, a multidisciplinary repository, managed by CERN in Geneva, which allows researchers to share and preserve research results in any size and form. Depositing data in ZENODO guarantees their compliance with the FAIR principles.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Rabinovich RA, Louvaris Z, Raste Y, Langer D, Van Remoortel H, Giavedoni S, Burtin C, Regueiro EM, Vogiatzis I, Hopkinson NS, Polkey MI, Wilson FJ, Macnee W, Westerterp KR, Troosters T; PROactive Consortium. Validity of physical activity monitors during daily life in patients with COPD. Eur Respir J. 2013 Nov;42(5):1205-15. doi: 10.1183/09031936.00134312. Epub 2013 Feb 8. PMID 23397303
- [Background] O'Hagen JM, Glanzman AM, McDermott MP, Ryan PA, Flickinger J, Quigley J, Riley S, Sanborn E, Irvine C, Martens WB, Annis C, Tawil R, Oskoui M, Darras BT, Finkel RS, De Vivo DC. An expanded version of the Hammersmith Functional Motor Scale for SMA II and III patients. Neuromuscul Disord. 2007 Oct;17(9-10):693-7. doi: 10.1016/j.nmd.2007.05.009. Epub 2007 Jul 19. PMID 17658255
- [Background] Berard C, Payan C, Hodgkinson I, Fermanian J; MFM Collaborative Study Group. A motor function measure for neuromuscular diseases. Construction and validation study. Neuromuscul Disord. 2005 Jul;15(7):463-70. doi: 10.1016/j.nmd.2005.03.004. PMID 16106528
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Erratum: ATS Statement: Guidelines for the Six-Minute Walk Test. Am J Respir Crit Care Med. 2016 May 15;193(10):1185. doi: 10.1164/rccm.19310erratum. No abstract available. PMID 27174486
- [Background] Mikolaizak AS, Rochester L, Maetzler W, Sharrack B, Demeyer H, Mazza C, Caulfield B, Garcia-Aymerich J, Vereijken B, Arnera V, Miller R, Piraino P, Ammour N, Gordon MF, Troosters T, Yarnall AJ, Alcock L, Gassner H, Winkler J, Klucken J, Schlenstedt C, Watz H, Kirsten AM, Vogiatzis I, Chynkiamis N, Hume E, Megaritis D, Nieuwboer A, Ginis P, Buckley E, Brittain G, Comi G, Leocani L, Helbostad JL, Johnsen LG, Taraldsen K, Blain H, Driss V, Frei A, Puhan MA, Polhemus A, Bosch de Basea M, Gimeno E, Hopkinson NS, Buttery SC, Hausdorff JM, Mirelman A, Evers J, Neatrour I, Singleton D, Schwickert L, Becker C, Jansen CP; clinical validation study (WP4) on behalf of Mobilise-D consortium. Connecting real-world digital mobility assessment to clinical outcomes for regulatory and clinical endorsement-the Mobilise-D study protocol. PLoS One. 2022 Oct 6;17(10):e0269615. doi: 10.1371/journal.pone.0269615. eCollection 2022. PMID 36201476
- [Background] Mazza C, Alcock L, Aminian K, Becker C, Bertuletti S, Bonci T, Brown P, Brozgol M, Buckley E, Carsin AE, Caruso M, Caulfield B, Cereatti A, Chiari L, Chynkiamis N, Ciravegna F, Del Din S, Eskofier B, Evers J, Garcia Aymerich J, Gazit E, Hansen C, Hausdorff JM, Helbostad JL, Hiden H, Hume E, Paraschiv-Ionescu A, Ireson N, Keogh A, Kirk C, Kluge F, Koch S, Kuderle A, Lanfranchi V, Maetzler W, Mico-Amigo ME, Mueller A, Neatrour I, Niessen M, Palmerini L, Pluimgraaff L, Reggi L, Salis F, Schwickert L, Scott K, Sharrack B, Sillen H, Singleton D, Soltani A, Taraldsen K, Ullrich M, Van Gelder L, Vereijken B, Vogiatzis I, Warmerdam E, Yarnall A, Rochester L. Technical validation of real-world monitoring of gait: a multicentric observational study. BMJ Open. 2021 Dec 2;11(12):e050785. doi: 10.1136/bmjopen-2021-050785. PMID 34857567
- [Background] Storm FA, Nair KPS, Clarke AJ, Van der Meulen JM, Mazza C. Free-living and laboratory gait characteristics in patients with multiple sclerosis. PLoS One. 2018 May 1;13(5):e0196463. doi: 10.1371/journal.pone.0196463. eCollection 2018. PMID 29715279
- [Background] Goldhahn J. Need for Digital Biomarkers in Musculoskeletal Trials. Digit Biomark. 2017 Aug 17;1(1):82-86. doi: 10.1159/000479753. eCollection 2017 Sep-Dec. PMID 32095748
- [Background] Stull DE, Leidy NK, Parasuraman B, Chassany O. Optimal recall periods for patient-reported outcomes: challenges and potential solutions. Curr Med Res Opin. 2009 Apr;25(4):929-42. doi: 10.1185/03007990902774765. PMID 19257798
- [Background] Leale I, Giustino V, Trapani P, Alonge P, Rini N, Cutro I, Leone O, Torrente A, Lupica A, Palma A, Roccella M, Brighina F, Di Stefano V, Battaglia G. Physical Activity in Patients with Neuromuscular Disease Three Years after COVID-19, a Longitudinal Survey: The After-Effects of the Quarantine and the Benefits of a Return to a Healthier Life-Style. J Clin Med. 2024 Jan 3;13(1):265. doi: 10.3390/jcm13010265. PMID 38202272
- [Background] Kennedy RA, Carroll K, McGinley JL, Paterson KL. Walking and weakness in children: a narrative review of gait and functional ambulation in paediatric neuromuscular disease. J Foot Ankle Res. 2020 Mar 2;13(1):10. doi: 10.1186/s13047-020-0378-2. PMID 32122377
- [Background] Retory Y, David P, Niedzialkowski P, de Picciotto C, Bonay M, Petitjean M. Gait Monitoring and Walk Distance Estimation With an Accelerometer During 6-Minute Walk Test. Respir Care. 2019 Aug;64(8):923-930. doi: 10.4187/respcare.06144. Epub 2019 Jun 18. PMID 31213569
- [Background] Ghislieri M, Gastaldi L, Pastorelli S, Tadano S, Agostini V. Wearable Inertial Sensors to Assess Standing Balance: A Systematic Review. Sensors (Basel). 2019 Sep 20;19(19):4075. doi: 10.3390/s19194075. PMID 31547181
- [Background] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966